CLINICAL TRIAL: NCT06634017
Title: Evaluation of Effect of Platelet-Rich Fibrin on Orthodontic Tooth Movement: a Split Mouth Randomised Controlled Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Fahad Iqbal Farooqui, Lecturer, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIFarooqui
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Rate of Tooth Movement in Orthodontic Patients

STUDY DESIGN:
Intervention Model Description: All routine history and medical records will be taken before commencing the treatment. The rate of orthodontic tooth movement and the root length of the canine will be measured using the calipers on cast model and the digital periapical X-Ray respectively using millimeter unit. All measurements will be recorded at the baseline (T0) followed by at the end of 8weeks (T1), before giving second dose of PRF, to assess single dose PRF outcomes and at end of 20 weeks (T2) to assess multiple dose PRF outcomes. Periapical x-rays to assess effect of single dose of PRF on root length will be taken at baseline (T0) just before injecting PRF and starting canine retraction and will be compared with the second periapical x-ray taken at the end of 8week (T1), just before injecting second dose of PRF.
Who Masked: Participant, Investigator
Masking Description: This trial will be a double-blind trial where the examiner and the patient both will be blind. Since the placebo and i-PRF will be in similar looking glass tubes the patient and the investigator/ examiner who is the orthodontist will not know which side of the maxilla has been intervened with i-PRF and which one with the placebo injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL (Experimental): Only the test side that will be intervened with i-PRF will be obtained from the upper liquid layer and will be placed in dental injectors using a 27 mm gauged needle. During the first application the amount of i-PRF will be standardized as 4 mL and injected through intra-ligamental into the disto-buccal and disto-palatal side of the canine tooth (2 mL for each side) and at the time of second intervention i.e 8th week form the baseline intramucosal injection will be administered equidistant from the maxillary canine and second premolar, 2ml on buccal side and 2ml on palatal side) after anesthetizing the region with local anesthesia (2% Lignocaine).
  Interventions: Biological: Platelet rich fibrin
- CONTROL (Placebo Comparator): On control side saline was injected using a 27 mm gauged needle. During the first application the saline was injected through intra-ligamental into the disto-buccal and disto-palatal side of the canine tooth (2 mL for each side) and at the time of second intervention i.e 8th week form the baseline intramucosal injection will be administered equidistant from the maxillary canine and second premolar, 2ml on buccal side and 2ml on palatal side) after anesthetizing the region with local anesthesia (2% Lignocaine).
  Interventions: Biological: Platelet rich fibrin

INTERVENTIONS:
Biological: Platelet rich fibrin — Only the test side that will be intervened with i-PRF will be obtained from the upper liquid layer and will be placed in dental injectors using a 27 mm gauged needle. During the first application the amount of i-PRF will be standardized as 4 mL and injected through intra-ligamental into the disto-buccal and disto-palatal side of the canine tooth (2 mL for each side) and at the time of second intervention i.e 8th week form the baseline intramucosal injection will be administered equidistant from the maxillary canine and second premolar, 2ml on buccal side and 2ml on palatal side) after anesthetizing the region with local anesthesia (2% Lignocaine).

SUMMARY:
it is a randomized control trial and aims at investigating the effects of PRF on rate of tooth movement and root length to be tested on larger sample size of pakistani population

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in the research
* Orthodontic patients with good oral hygiene
* Patients with periodontal probing depths≤3 mm with no bone loss
* Patients undergoing orthodontic treatment with fixed appliance and requiring upper first premolar extraction followed by canine retraction
* Patients treated with canine retraction utilizing maximum anchorage in the maxillary arch from trans-palatal arch anchorage device
* Patients with mild to moderate crowding in maxillary arch
* Patients with no previous history of orthodontic treatment

Exclusion Criteria:

* patients who are smokers, health compromised (such as diabetics, with bone disorders, immunocompromised, known with blood dyscrasias) will be excluded from the trial. Patients with drug history of non-steroidal anti-inflammatory drugs, anti-inflammatory (in last 30 days), antibiotic therapy in last 3 months and those women who are pregnant will also be excluded.

Other exclusion criteria will be patients with hypodontia, impacted/ectopic canines, extracted first molars, and patients who may discontinue the trial with or without assigning any reasons and those not consenting to participate in the research.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
: Distance of canine retraction in millimeters / month in different groups-control, single dose PRF and multiple doses of PRF. | 5 months

SECONDARY OUTCOMES:
Difference in root length of canine measured before and after canine retraction and compared amongst different groups | 5 month

CONTACTS AND LOCATIONS:
Locations (1):
- Dow university of health sciences, Karachi, Sindh, Pakistan